CLINICAL TRIAL: NCT00459823
Title: A Phase I Open-Label, Single-Arm, Dose Escalation Study of E7107 Administered IV (Bolus) on Days 1, 8, and 15 Every 28 Days to Patients With Solid Tumours
Brief Title: A Dose Escalation Study of E7107 Administered IV (Bolus) on Days 1, 8, and 15 Every 28 Days to Patients With Solid Tumours
Status: Suspended | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Limited (Industry)
Responsible Party: Eisai Limited Medical Information Services, Eisai Limited
Organization: Eisai Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E7107-E044-102
Record Dates: First submitted 2007-04-11; First posted 2007-04-13 (Estimated); Last update posted 2009-03-24 (Estimated); Status verified 2009-03

CONDITIONS: Cancer
Keywords: Cancer; solid tumors
MeSH Terms: conditions — Neoplasms | interventions — E 7107

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: E7107

INTERVENTIONS:
Drug: E7107 — E7107 administered by intravenous infusion (as a 2-5 minutes bolus) on days 1, 8 and 15 every 28 days.

SUMMARY:
Two-centre, open-label, non-randomized, dose-finding phase I study to determine the MTD of E7107 administered by intravenous infusion (as a 2-5 minutes bolus) on days 1, 8 and 15 every 28 days in patients with solid tumors, for whom therapy of proven efficacy does not exist or is not longer effective.

ELIGIBILITY:
INCLUSION CRITERIA:

Patients must meet all of the inclusion criteria outlined below in order to be eligible to participate in the study.

1. Patients with histologically and/or cytologically confirmed solid tumours who have progressed after receiving approved therapies for their disease and for whom no curative therapies are available.
2. Surgery and radiotherapy must have been completed at least four weeks prior to study entry, and prior chemotherapy and other anti-cancer therapy, excluding bisphosphonates at a steady dose level, must have been discontinued for at least two weeks previously. All acute toxicities related to these treatments must have resolved.
3. Aged >= 18 years.
4. ECOG performance status score of 0 or 1.
5. Written informed consent prior to any study specific screening procedures, which will include voluntary additional consent to provide specimens specifically for pharmacogenomic analysis, with the understanding that the patient may withdraw consent at any time without prejudice.
6. Willing and able to comply with the protocol for the duration of the study.
7. Anticipated life expectancy > three months.
8. After MTD has been reached: patients must have measurable disease according to RECIST criteria.

EXCLUSION CRITERIA:

Patients with the following characteristics will not be eligible for the study:

1. Symptomatic or progressive brain tumours or brain or leptomeningeal (CNS) metastases requiring clinical intervention, except if they have completed local therapy and have discontinued the use of corticosteroids for this indication for at least two weeks before starting treatment with E7107.
2. Any of the following laboratory parameters:

   1. haemoglobin < 9 g/dL (5.6 mM)
   2. neutrophils <1.5 x 10^9/L
   3. platelets <100 x 10^9/L
   4. serum bilirubin >25 ìM (1.5 mg/dL)
   5. liver function tests (defined as AST and ALT) with values >3 x ULN (5 x ULN if liver metastases are present)
   6. serum creatinine > 105µM (or >1.5 mg/L) or creatinine clearance < 40 mL/min
3. Positive history of HIV, active hepatitis B or active hepatitis C or severe/uncontrolled intercurrent illness or infection.
4. Clinically significant cardiac impairment or unstable ischemic heart disease (greater than Class III according to NYHA classification) including a myocardial infarction within six months of study start.
5. Bleeding or thrombotic disorders, or using therapeutic dosages of anticoagulants.
6. History of alcoholism, drug addiction, or any psychiatric or psychological condition which, in the opinion of the Investigator, would impair study compliance.
7. Pregnancy or lactation (all women of childbearing potential must have a negative pregnancy test before inclusion in the study; peri-menopausal women must have been amenorrheic for at least 12 months, otherwise pregnancy test is required).
8. Fertile persons who are not willing to use adequate contraception (defined as two forms of contraception including a barrier method).
9. Patients with a marked screening or baseline prolongation of QT/QTc interval (i.e., repeated demonstration of a QTc interval > 450 msec); a history of additional factors of TdP (i.e., heart failure, hypokalaemia, family history of Long QT Syndrome).
10. Legal incapacity.
11. After MTD has been reached: Second malignancy within the past 5 years, except for carcinoma in situ of the cervix, basal cell carcinoma of the skin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2007-05; Primary Completion 2009-06 (Estimated)

PRIMARY OUTCOMES:
To determine MTD of E7107. Safety and tolerability. | Every six weeks.

SECONDARY OUTCOMES:
Pharmacokinetics of E7107. Evaluation of anti-tumor activity. To investigate potential biomarkers of pharmacodynamic effect. | Every 21 days.

CONTACTS AND LOCATIONS:
Overall Officials: Jantien Wanders, M.D., Study Director — Eisai Limited
Locations (2):
- Department of Medical Oncology, Erasmus University Medical Centre, Rotterdam, Netherlands
- Medical Oncology Service. Vall d'Hebron University Hospital, Barcelona, Spain